CLINICAL TRIAL: NCT04574726
Title: Study of Balance Reactions in a Virtual Environment Compared to a Real Environment
Acronym: EQUIVIRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pôle Saint Hélier (Other)
Collaborators: Hopital La Musse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 2020-A01841-38
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, controlled, randomized, intervention study with minimal risks and constraints (RIPH2) on healthy volunteers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual environment (Experimental): Balance test in virtual environment with a virtual reality software executed in a 6DOF Occulus Quest helmet and a motion capture software with a Kinect Azure DK camera.
  Interventions: Other: static balance; Other: dynamic balance
- reel environment (Active Comparator): Balance test in real environment with a motion capture software and a Kinect Azure DK camera.
  Interventions: Other: static balance; Other: dynamic balance

INTERVENTIONS:
Other: static balance — 30-second right and left unipodal static balance test
Other: dynamic balance — for the unipodal dynamic balance test, 4 movements will be done by the volunteers in this order :
  * 180° elevation of the arms
  * lowering of the arms on the side of the single-legged support to the horizontal position
  * 180° horizontal translation of the arms
  * return from the horizontal to the starting point

SUMMARY:
Validate a virtual environment by demonstrating a non modification of the characteristics of postural reaction and displacement of the body's center of pressure between a real environment and the same environment in immersive virtual reality.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer, men and women over 18 years old

Exclusion Criteria:

* Severe visual disorders which couldn't enable immersive virtual reality experience
* Immobilisation of one of the upper limbs (restraint splint)
* Orthopedic problems and pain in the lower limb
* MSSQ upper than 25
* Pregnant women
* Person under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Area of CoP (Center of pression) | Immediately after inclusion
  Mesure of area of center of pression during the balance tests in virtual condition and real condition, order in terms of randomisation

SECONDARY OUTCOMES:
Total distance covered by the CoP during the balance test (in mm) | Immediately after inclusion
  Mesure of the total distance covered by the CoP during the balance tests (in mm) in virtual condition and real condition, order in terms of randomisation
Simulator Sickness Quantifying (SSQ) | Immediately after the balance test
  SSQ completed after the balance test, SSQ is a scale of cyber sickness, from 0 to 48.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Pole Saint-Hélier, Rennes, Brittany Region
  - Hôpital la Musse, Saint-Sébastien-de-Morsent

IPD SHARING:
Plan to Share IPD: Undecided